CLINICAL TRIAL: NCT04728048
Title: A Randomized Clinical Study to Compare the Number of Physician Top-up Interventions During the First Stage of Labour Between Two Different Neuraxial Analgesia Techniques: the Dural Puncture Epidural and the Standard Epidural
Brief Title: Dural Puncture Epidural VS Standard Epidural on Physician Top-ups During Labour Analgesia
Acronym: DPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Principal Investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-2334
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Obstetric Pain; Labor Pain; Anesthesia
Keywords: Dural puncture epidural; Epidural; Low dose bupivacaine
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural puncture epidural (group DPE) (Experimental): The epidural space will be identified in the seated position between the L2 and L5 interspaces with a 17G-10 cm Tuohy epidural needle (CHS ®, Oakville, ON, Canada) using a loss of resistance to saline technique. In both groups, a needle-through-needle technique will be performed using a 25G 5-inch Whitacre spinal needle (BD®, Franklin Lakes, NJ, USA). In group DPE, a single dural puncture with confirmation of free-flow CSF will be performed. If there is no free-flow CSF return through the spinal needle, the epidural catheter will be threaded 4-5cm in the epidural space and the patient will still be assigned to the DPE group, as per "intent-to-treat" protocol.
  Interventions: Procedure: Dural puncture epidural
- Standard epidural (group EPL) (Active Comparator): The epidural space will be identified in the seated position between the L2 and L5 interspaces with a 17G-10 cm Tuohy epidural needle (CHS ®, Oakville, ON, Canada) using a loss of resistance to saline technique. In both groups, a needle-through-needle technique will be performed using a 25G 5-inch Whitacre spinal needle (BD®, Franklin Lakes, NJ, USA).In Group EPL, no dural puncture will be performed and the catheter will be threaded 4-5cm in the epidural space.
  Interventions: Procedure: Standard epidural

INTERVENTIONS:
Procedure: Dural puncture epidural — already described
  Arms: Dural puncture epidural (group DPE)
Procedure: Standard epidural — already described
  Arms: Standard epidural (group EPL)

SUMMARY:
The purpose of this prospective randomized controlled study is to compare the number of physician top-up interventions during the first stage of labour between two different neuraxial analgesia techniques : the dural puncture epidural and the standard epidural.

DETAILED DESCRIPTION:
Providing adequate labour analgesia has always been an important issue in obstetrical anesthesia. Different types of neuraxial techniques include standard epidural analgesia (EPL), combined spinal epidural analgesia (CSE) and dural puncture epidural analgesia (DPE). DPE, which has gained in popularity in recent years, is similar to CSE in which the dura mater is punctured, however without injection of medication in the cerebrospinal fluid (CSF). Recent studies have found benefits of the DPE technique, such as less fetal bradycardia than CSE, better bilateral sacral analgesia than EPL and faster onset than EPL. No study has yet compared DPE to EPL when an ultra-low concentration of local anesthetic protocol is used for maintenance of analgesia. We hypothesize that in term primiparous and multiparous parturients, a dural puncture epidural technique will improve labour analgesia quality during the first stage of labour (based on physician top-up interventions) compared with a standard epidural technique when a patient-controlled epidural analgesia (PCEA) with ultra-low concentration epidural mixture classically used in our institution based on our hospital orders and national guidelines.

The main hypothesis for this study is to show that there will be 50% reduction in the incidence of parturients in need of at least one physician top-up intervention during the first stage of labour in the DPE group compared to the EPL group.

The patients will be approached by the anesthesia research team upon arrival at the birth unit. The randomization will be done at the time the parturient requests an epidural. Randomization will be done in a 1:1 ratio until we reach 65 subjects in each group.

Before neuraxial catheter placement, a 20G or 18G intravenous (IV) catheter is inserted and standard monitoring is applied.

The attending or resident in anesthesiology will place the neuraxial catheter following the next steps :

* Epidural space is identified in seated position (L2-L3 or L3-L4) using an epidural needle 17G 10 cm Tuohy.
* Loss of resistance to saline technique.
* In both groups, a needle-through-needle technique is performed using a 25G 5-inch Whitacre spinal needle.
* In group DPE, a single dural puncture with confirmation of free-flow CSF is performed and in group EPL no dural puncture is performed.
* Catheter is placed 4-5 cm in the epidural space: 19G multi-orifice Perifix FX catheter.

Initiation of analgesia in both groups will be as followed :

* Test dose of 3mL bupivacaine 0,25%.
* Initial bolus (10mL Bupivacaine 0,125% plus fentanyl 50mcg) fractioned in two doses.
* PCEA is then initiated with a basal infusion of 6mL/h (solution of bupivacaine 0,0625% + fentanyl 2mcg/mL) and 8 mL boluses are permitted every 20 minutes.

If analgesia is inadequate, defined as NPRS ≥ 4, within the first 30 minutes of epidural initiation OR more than 30 minutes after catheter placement and after 2 PCEA boluses in less than 1 hour, the initial step will be to administered a nurse top-up intervention: 10 mL bolus of the epidural infusion (bupivacaine 0,0625% + fentanyl 2mcg/mL) via the infusion pump. If analgesia is still inadequate 30 minutes after initial nurse top-up intervention, the anesthesiologist is called, the catheter is pulled back 1cm and a physician manual top-up 10mL bolus of bupivacaine 0,125% is administered. If 30 minutes after the physician manual top-up bolus analgesia is still inadequate, analgesia management is transferred to the attending anesthesiologist.

Standard nurse care during and after catheter placement will be applied following an already established protocol at our center.

Analgesia will be evaluated using the verbal NPRS from Gélinas C. (2007) that allows parturients to rate their pain on a scale from 0 to 10. Sensory blockade will be evaluated using ice. The evaluation will start at the S2 dermatome, where S2 is assessed at the midpoint of the popliteal fossa, and will be moving in a caudad to cephalad direction. The evaluator will assess asymmetrical blockade, which is defined as a difference in sensory blockade to cold sensation greater than 2 dermatomal levels between the left and right side of the patient. Motor blockade will be evaluated using the Bromage score (1978).

Ambulation criteria will be evaluated at certain times following initial physician bolus. The criteria already established in our center are listed below:

* No obstetrical contraindications.
* Sensory blockade ≤ T4.
* Absence of motor blockade according to Bromage score (score = 4).
* Systolic blood pressure ≥ 90 mmHg AND/OR a fall of less than 20 mmHg compared to the patient's initial systolic blood pressure.
* Negative postural hypotension test.
* Successful squat test.

Parturients overall satisfaction with neuraxial analgesia will be evaluated the day following delivery. Presence or absence of post dural puncture headache symptoms will be noted at 24h post partum.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women (ASA 1 and 2) requesting epidural analgesia during labour.
2. Primiparous and multiparous parturients at term gestation (37 to 42 weeks).
3. Women 18 years old and older.
4. Administration of epidural analgesia between 7am and 4pm on weekdays.
5. Singleton and vertex presentation foetus.
6. Cervical dilatation ≤ 5 cm.
7. BMI ≤ 40.
8. French speaking

Exclusion Criteria:

1. Pregnancy diseases such as gestational hypertension, preeclampsia and gestational diabetes.
2. Contraindications to neuraxial analgesia: thrombocytopenia < 70 x 109/L, spinal cord anomalies, anticoagulation therapy, etc.
3. Known important fetal anomalies.
4. Allergy to any of the medications used in the study.
5. Suspected chorioamnionitis with spontaneous premature rupture of membranes (PROM).
6. Difficulty understanding and speaking French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Need for 1 physician epidural top-up | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  The number of parturients who need at least one physician top-up intervention during the first stage of labour.

SECONDARY OUTCOMES:
Number of physician epidural top-ups | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To compare the number of physician top-up interventions necessary in the first stage of labour between both groups.
Timing of physician top-ups | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To measure the timing of request for physician top-up interventions and timing of actual physician top-up interventions.
Analgesia scores | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To evaluate the analgesia, using the verbal numeric pain rating scale (NPRS) from 0 to 10, every 5 minutes after catheter placement until NPRS ≤ 3, and then every hour. Each time, the parturient will evaluate her maximal pain during the last contraction. If the parturient is sleeping and does not wake up in the 30 minutes following the planned analgesia evaluation, we will respect sleep and consider that the analgesia is adequate at that time and will be scored at 0 on the NPRS.
Sacral block | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To assess the incidence of S2 bilateral blockade every hour, where S2 is assessed at the midpoint of the popliteal fossa.
Asymetrical block | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To assess the incidence of asymmetrical blockade every hour, which is defined as a difference in sensory blockade to cold sensation greater than 2 dermatomal levels between the left and right sides of the patient.
Motor block | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To assess the presence of motor blockade every hour, using the Bromage score (1 to 4).
Ambulation criteria | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To determine the number of parturients that fulfill ambulation criteria at 30 min, 1 hour and 2 hours after catheter placement.
Ambulation | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To determine the number of parturients that ambulate at any moment during the first stage of labour.
Urinary catheterisation | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To determine the number of parturients who need urinary catheterisation for any indication.
Local anesthetic and fentanyl doses | Up to 24 hours after inclusion. From installation of epidural analgesia until the end of first stage of labour defined as full cervix dilation or decision by the attending obstetrician to proceed to a cesarean delivery.
  To determine the total quantity of local anesthetic (mg) and fentanyl (mcg) that are received during the first stage labour in both groups, including the top-up boluses.
Patient satisfaction | Up to 48 hours after inclusion.
  To evaluate the parturients overall satisfaction with neuraxial analgesia 24 hours postpartum, using a 0 to 100 scale. A cutoff of ≤ 60 will be taken as poor satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Île de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No